CLINICAL TRIAL: NCT07061626
Title: A Two-Part, Phase 1/2a Trial to Determine the Maximum Tolerated Dose, Safety, and Tolerability of Rhenium (186Re) Obisbemeda (Rhenium-186 NanoLiposome, 186RNL) Delivered Via Convection Enhanced Delivery (CED) in Supratentorial Recurrent, Refractory, or Progressive Pediatric Ependymoma and High-Grade Glioma (HGG)
Brief Title: Determine Maximum Tolerated Dose, Safety, and Tolerability of Rhenium (186Re) in Pediatric Recurrent, Refractory or Progressive Ependymoma and High-Grade Glioma
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Plus Therapeutics (Industry)
Collaborators: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CA-2024-PBC-001; HT9425-24-1-1035 (Other Grant/Funding Number: Department of Defense Congressionally Directed Medical Research Program)
Record Dates: First submitted 2025-05-03; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Ependymoma; High Grade Gliomas
MeSH Terms: conditions — Ependymoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1a - Cohort A (Experimental): Up to six subjects will be enrolled in Cohort A. Tumor size will be limited to a maximum diameter of (less than or equal to) ≤2 cm and a maximum volume of (less than or equal to) ≤4.2 mL. Up to two CED catheters will be utilized in Cohort A at the discretion and consensus of the PI, neurosurgeon, and/or study team. The concentration of 186RNL infusate in Cohort A is 0.5 mCi/mL, with a corresponding estimated absorbed dose of ~87.5Gy.
  Interventions: Drug: Rhenium-186 Nanoliposome
- Phase 1a - Cohort B (Experimental): Up to six subjects will be enrolled in Cohort B. Tumor size will be limited to a maximum diameter of 3.5 cm in the longest axis and a maximum volume of 22.4 mL. Up to 5 total catheters may be used for Cohort B at the discretion and consensus of the PI, neurosurgeon, and/or study team to ensure total tumor volume coverage. The concentration of 186RNL infusate in Cohort B is 1.0 mCi/mL with a corresponding estimated absorbed dose of ~176Gy (~2x Cohort A).
  Interventions: Drug: Rhenium-186 Nanoliposome
- Phase 1b (Experimental): Phase 1b continued dosing escalation will be defined following review of the safety data from Phase 1a.
  Interventions: Drug: Rhenium-186 Nanoliposome
- Phase 2 (Experimental): The Phase 2 expansion study will utilize the maximum tolerable dose (MFD) determined from the Phase 1 dose escalation study. If no maximal tolerable dose is found, tumors may be treated up to an estimated total absorbed dose of 176 Gy. Varying concentrations of 186RNL infusate (0.5-2.5 mCi/mL) may be used to achieve this maximum tolerable dose while maintaining total tumor volume coverage. Phase 2a will enroll an additional 12 patients with a diagnosis of recurrent, refractory, or progressive ependymoma and an additional 20 patients with a diagnosis of recurrent, refractory, or progressive HGG.
  Interventions: Drug: Rhenium-186 Nanoliposome

INTERVENTIONS:
Drug: Rhenium-186 Nanoliposome — Rhenium (186Re) Obisbemeda (Rhenium-186 NanoLiposome, 186RNL), BMEDA-chelated-186rhenium encapsulated within liposomes, allows the 186Re to be directly delivered to the site of the tumor through CED and maintain localization at the site of infusion.

SUMMARY:
Pediatric patients 6-21 years of age with supratentorial recurrent, refractory, or progressive pediatric ependymoma and high-grade glioma (HGG) will be included in this study of treatment with Rhenium-186 Nanoliposome (186RNL). Phase 1 of the study will look to determine the maximum tolerated dose (MTD) of 186RNL in this patient population. Phase 2 of the study will use the recommended dose determined in Phase 1 to continue to look at overall response rate and progression-free survival following 186RNL treatment.

ELIGIBILITY:
Inclusion Criteria:

1. 6 years to 21 years* of age.
2. Lesion number and size:

   1. Phase 1a/b only: A single lesion (less than or equal to) ≤3.5 cm (longest axis) and volume of (less than or equal to) ≤22.4 mL as the largest tumor (subsequent to individual Cohort lesion size requirements).
   2. Phase 2a only: A single lesion or any number of multiple lesions separated by (less than or equal to) ≤3 cm; each lesion (less than or equal to) ≤3.5 cm (longest axis) and volume of (less than or equal to) ≤22.4 mL as the largest tumor.
3. Diagnosis:

   a) Documented recurrent, refractory, or progressive ependymoma or HGG not eligible for resection or no longer receiving standard of care.

   i) Phase 2a only: May include patients with recurrent, refractory, or progressive ependymoma or HGG where SOC surgery could be safely delayed four (4) weeks post-infusate.

   b) Documented histologically confirmed high-grade glioma [following 2021 WHO CNS5 glioma nomenclature, e.g., Anaplastic astrocytoma, Anaplastic pleomorphic xanthoastrocytoma (PXA), Anaplastic ganglioglioma, Anaplastic oligodendroglioma, Glioblastoma, Diffuse midline glioma, H3K27M mutant].
4. Karnofsky Performance Status ≥ 60. For subjects <16 years of age, Lansky score ≥ 60.
5. Acceptable liver function:

   1. Bilirubin ≤ 1.5 times the upper limit of normal
   2. AST (SGOT) and ALT (SGPT) ≤ 3.0 times the upper limit of normal (ULN)

      6) Acceptable renal function:

   <!-- -->

   1. Serum creatinine ≤1.5xULN

7. Acceptable hematologic status (without hematologic support):

1. ANC ≥1000 cells/uL
2. Platelet count ≥100,000/uL
3. Hemoglobin ≥9.0 g/dL

   8. All subjects of childbearing potential must have a negative serum pregnancy test, and subjects must agree to use effective means of contraception (for example, surgical sterilization or the use of barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel or an IUD) with their partner from entry into the study through 6 months after the last dose.

   9. Life expectancy of at least 2 months.

   *Will consider treatment of subjects up to 25 years of age on a per-patient basis if no other co-morbidities are present that require subspecialty consultation outside of neurosurgical and oncologic care.

Exclusion Criteria:

1. Spinal disease.
2. Infratentorial location of tumor.
3. Involvement of the leptomeninges.
4. Serious intercurrent illness, as determined by the treating physician, which would compromise either patient safety or study outcomes such as:

   1. Hypertension (two or more blood pressure readings performed at screening of systolic blood pressure (SBP) or diastolic blood pressure (DBP) above 95th percentile for age) despite optimal treatment.
   2. Active medically significant infection unresponsive to antibiotics (e.g., non-healing wound, ulcer), uncontrolled systemic infection, or bone fracture.
   3. Clinically significant cardiac arrhythmias.
   4. Untreated hypothyroidism.
   5. Congestive heart failure.
   6. Myocarditis.
   7. Inherited bleeding diathesis or coagulopathy with the risk of bleeding.
   8. Known active malignancy other than ependymoma or high-grade glioma.
5. Any of the following prior anticancer therapy:

   1. Prior treatment with Bevacizumab or other VEGF agents within 12 months prior to study registration.
   2. Non-standard radiation therapy such as brachytherapy, systemic radioisotope therapy, or intra-operative radiotherapy (IORT) to the target site at any time prior to study registration.
   3. Standard radiation therapy within 12 weeks prior to study registration.
   4. Any systemic therapy within 28 days or 2 half-lives, whichever is longer, prior to study registration (this may include investigational agents, small-molecule kinase inhibitors, non-cytotoxic hormonal therapy, biologic agents, metronomic/protracted low-dose chemotherapy, etc.).
   5. Nitrosoureas or mitomycin C within 42 days prior to study registration.
6. Psychiatric illness/social situations that would limit compliance with the study requirements.
7. A tumor located within 1.0cm of a ventricle AND it is determined by the surgeon, PI, and Sponsor to be a risk for drug extravasation to the subarachnoid space if given catheter placement and drug administration.
8. A tumor within 1.5cm of critical structures, including the optic chiasm, optic nerves, or brainstem.
9. Evidence of acute intracranial or intratumoral hemorrhage either by magnetic resonance imaging (MRI) or computerized tomography (CT) scan (subjects with resolving hemorrhage changes, punctate hemorrhage, or hemosiderin are eligible).
10. Treatment with antiepileptic medications must have a two-week history of a stable dose of antiepileptic without seizures prior to study registration.
11. Patients with corticosteroid requirements to control cerebral edema must be maintained at a stable or decreasing dose for a minimum of two weeks without progression of clinical symptoms prior to study registration.

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 28 days
  Determine the maximum tolerated dose (MTD) of 186RNL administered by convection-enhanced delivery (CED) in subjects with supratentorial recurrent, refractory, or progressive pediatric ependymoma or HGG.
Overall Response Rate (ORR) by RANO in Ependymoma | 90 days
  Determine the best overall response rate (ORR) by Radiographic Assessment in Neuro-Oncology (RANO) criteria following 186RNL administration in subjects with supratentorial recurrent, refractory, or progressive pediatric ependymoma.
Progression-Free Suvival at 12 months (PFS12) in HGG | 12 months
  Determine progression-free survival at 12 months (PFS12) in subjects with supratentorial recurrent, refractory, or progressive pediatric HGG.

SECONDARY OUTCOMES:
Safety of 186RNL Dose | 28 days
  Assess the safety of single dose 186RNL administered by CED in subjects with supratentorial recurrent, refractory, or progressive pediatric ependymoma or HGG, as determined by the most recent version of the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE).
Dose Distribution of 186RNL | 8 days
  Assess the dose distribution of 186RNL administered by CED in subjects with supratentorial recurrent, refractory, or progressive pediatric ependymoma or HGG.
Neuropsychologic Outcome | 1 year
  Assess the neuropsychologic outcomes of subjects exposed to 186RNL at 1 year in subjects with supratentorial recurrent, refractory, or progressive pediatric ependymoma or HGG using the following assessments. Wechsler Intelligence Scale for Children, Fifth Edition (WISC-V; ages 6-16:11) OR Wechsler Adult Intelligence Scale, Fourth Edition (WAIS-5; age >17): Vocabulary, Block Design, Symbol Search, Coding, Digit Span California Verbal Learning Test, Children's Version (CVLT-C; ages 6-16:11) OR California Verbal Learning Test, Third Edition (CVLT-3; age >17) Wide Range Assessment of Memory & Learning, Third Edition (WRAML3; all ages): Story Memory, Design Learning Beery-Buktenica Developmental Test of Visual-Motor Integration (Beery VMI; all ages)
Progression-Free Survival at 24 Months (PFS24) in Ependymoma | 24 months
  Determine the progression-free survival at 24 months (PFS24) in subjects with supratentorial recurrent, refractory, or progressive pediatric ependymoma.
Overall Response Rate (ORR) by RANO in HGG | 90 days
  Determine the best overall response rate (ORR) by Radiographic Assessment in Neuro-Oncology (RANO) criteria following 186RNL administration in subjects with supratentorial recurrent, refractory, or progressive pediatric HGG.
Overall Survival at 24 Months (OS24) | 24 months
  Determine overall survival at 24 months (OS24) in participants with supratentorial recurrent, refractory, or progressive pediatric ependymoma and in participants with supratentorial recurrent, refractory, or progressive pediatric HGG.

OTHER OUTCOMES:
Overall Response Rate (ORR) by RAPNO | 90 days
  Assess overall response rate (ORR) by Response Assessment in Pediatric Neuro-Oncology (RAPNO).
Tissue Sample from Standard of Care Surgical Resection of Tumor | 28 days
  In Phase 2a only: tissue sample collected from SOC surgical resection of tumor for microscopic activity 4 weeks after receiving treatment.